CLINICAL TRIAL: NCT05686993
Title: Effect of a Proposed Cav1.3 Inhibitor in Primary Aldosteronism - a Pilot Study
Brief Title: Effect of a Proposed Cav1.3 Inhibitor in Primary Aldosteronism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 154739
Record Dates: First submitted 2022-12-22; First posted 2023-01-17 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Primary Aldosteronism; Endocrine Hypertension
Keywords: Primary aldosteronism; Calcium channel blocker; Aldosterone
MeSH Terms: conditions — Hyperaldosteronism | interventions — Cinnarizine; cynarine; Nifedipine

STUDY DESIGN:
Intervention Model Description: Treatment with 2 study drugs with 2 weeks of drug washout in between Study drug treatments are: cinnarizine for 2 weeks, nifedipine for 2 weeks Order randomly determined by computer program, with results released by an independent clinician as patients are recruited
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cinnarizine and nifedipine (Experimental): Drug 1 for 2 weeks, 2 weeks of washout, then Drug 2 for 2 weeks Drug 1 and 2, in no specified order, Cinnarizine 30 mg oral TDS and Nifedipine 60 mg oral daily
  Interventions: Drug: Cinnarizine; Drug: NIFEdipine ER

INTERVENTIONS:
Drug: Cinnarizine — Cinnarizine oral 30mg TDS
  Other Names: Stugeron, Stunarone, Cinarin
Drug: NIFEdipine ER — Nifedipine oral 60mg daily extended release
  Other Names: Adalat, Adipine, Coracten, Fortipine, Nifedipress

SUMMARY:
The goal of this pilot, open-label prospective study is to evaluate if the effect of calcium channel blockade on plasma aldosterone levels in people with primary aldosteronism (PA) is due primarily to Cav1.3 blockade.

This will be tested by treating participants who have PA with both cinnarizine (Cav1.3 blocker) and nifedipine (Cav1.2 blocker) and evaluating effect on aldosterone levels and blood pressure over a two week course of treatment.

DETAILED DESCRIPTION:
Medical treatment for Primary Aldosteronism (PA) is currently limited to mineralocorticoid receptor antagonists (MRA), the most widely available of which is spironolactone. This can cause numerous adverse effects, especially in men, due to interference with androgen and progesterone signalling. Hence, alternative drug targets are needed, one potential of which is Cav1.3.

The CACNA1D mutation in PA affects the calcium channel Cav1.3. Cav1.3 inhibition may offer targeted treatment for patients with mutations in CACNA1D. Cav1.3 has been a candidate for novel inhibitors of aldosterone production,4 for which the case is enhanced if CACNA1D-mutations underlie the above-described phenotype of PA (asymmetric disease leading to failure to achieve cure with adrenalectomy).

The calcium-channel blocker, cinnarizine, typically used for vertigo and nausea, has been identified to fit the recently described crystal structure of Cav1.3. This raises the possibility of using this drug to assess the effect of Cav1.3 inhibition in PA. This may lead to further studies involving randomisation and placebo to determine if Cav1.3 inhibition is an important method by which aldosterone levels can be lowered in people with PA.

This study seeks to explore whether the effect of calcium channel blockade on aldosterone levels in people with PA is due to Cav1.3 blockade, by comparing cinnarizine (proposed Cav1.3 inhibitor) to a conventional calcium channel blocker nifedipine (Cav1.2 inhibitor). Cinnarizine is not a likely prospect for long-term treatment of PA, because of its potential additional actions as well as Cav1.3 blockade, but using it in this setting, for a short period of time, allows exploration of a property of this existing drug (Cav1.3 inhibition). Outcomes could form the basis of further exploration of this mechanism for future PA treatments.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed PA, as demonstrated by a positive screening test and internationally endorsed confirmatory test (saline suppression test, captopril challenge test)
* Adults > 18 years of age
* Able and willing to give informed consent

Exclusion Criteria:

* Uncontrolled hypertension requiring use of MRA
* Unwilling or unable to give consent
* Below age 18 or above age 90 years
* Allergy to cinnarizine or nifedipine or their excipients
* Existing use of cinnarizine or nifedipine for an alternative indication
* Breastfeeding or pregnant women
* Diagnosis of Parkinson's disease
* Severe hepatic or renal insufficiency
* Concurrent use of sedating central nervous system (CNS) depressants or rifampicin
* Porphyria
* Cardiogenic shock, clinically significant aortic stenosis, unstable angina, within one month of a myocardial infarction
* Previous gastro-intestinal or oesophageal obstruction or ileostomy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-04-24 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-06 (Actual)

PRIMARY OUTCOMES:
Aldosterone change | 6 weeks
  Evaluate whether the effect of calcium channel blockade on plasma aldosterone levels is due primarily to Cav1.3 blockade in individuals with PA and clinical features suggesting an increased likelihood of a CACNA1D mutation.

SECONDARY OUTCOMES:
Blood pressure change | 6 weeks
  Evaluate whether the use of a proposed Cav1.3 inhibitor affects blood pressure in individuals with PA, evaluating both systolic blood pressure and diastolic blood pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Morris Brown, MD FRCP, Principal Investigator — Queen Mary University of London
Locations (1):
- St Bartholomew's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ng E, Lee YN, Taylor A, Shaheen F, Azizan E, Drake WM, Brown MJ. Evaluation of Aldosterone Suppression by Cinnarizine, a Putative Cav1.3 Inhibitor. J Clin Endocrinol Metab. 2025 Sep 16;110(10):2752-2761. doi: 10.1210/clinem/dgaf081. PMID 40052842